CLINICAL TRIAL: NCT05288647
Title: Efficacy of Computer-guided Versus Conventional Sodium Hyaluronate Injection in Superior Joint Space in Treatment of Intra-articular TMJ Disorder
Brief Title: Computer Guided Versus Conventional TMJ Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, AbdElKader Ahmed Hyder Mohamed, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CG-HA-TMJ-inj.
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: TMD
Keywords: TMD

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Patients treated with four computer-guided sodium hyaluronate injections in superior TMJ space.
  Interventions: Procedure: TMJ injection
- Group B (Active Comparator): Patients treated with four conventional sodium hyaluronate injections in superior TMJ space.
  Interventions: Procedure: TMJ injection

INTERVENTIONS:
Procedure: TMJ injection — four sodium hyaluronate injections in superior TMJ space

SUMMARY:
This study is designed to evaluate the clinical outcomes of computer-guided sodium hyaluronate injection in superior joint space in comparison to conventional injection for treatment of intra-articular TMJ disorder.

DETAILED DESCRIPTION:
This study aimed to reveal the superiority of computer-guided TMJ injection (if found) above the conventional method from the clinician and patient point of view.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with intra-articular TMJ disorder according to Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD).
* Patients who would not respond to conservative treatment as the first line of treatment.

Exclusion Criteria:

* Patients with polyarthritis or degenerative joint disease.
* Patients with myofascial pain.
* Previous history of minimally invasive or invasive treatment of TMJ.
* History of mandibular fracture.
* Lactating, pregnant or planning pregnancy women.
* Known hypersensitivity to hyaluronic acid or clear biocompatible photopolymer resin.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
Comparison of maximum unassisted mouth opening range | 6 months
  Opening range determined by asking the patient to gently open the mouth and measure the distance between upper and lower central incisor using an vernier digital electronic caliper. Vertical movement of the mandible corrected by adding the vertical overlap.
Comparison of modified Helkimo's clinical dysfunction index. | 6 months
  A modified version of Helkimo's clinical dysfunction index calculated to assess the TMJ dysfunction.
Comparison of pain intensity on Visual analog scale | 6 months
  Patients asked to mark their TMJ-related pain level on a scale from 0 to 10, where 0 is "no pain" and 10 is "severe pain".

SECONDARY OUTCOMES:
Total procedural time. | Baseline
  Total procedural time consumed starting from application of topical antiseptic up to the end of the procedure.
Patient convenience. | Baseline
  Patient convenience on a scale from "0" to "10", where "0" is highly convenient and "10" extremely intolerable.

CONTACTS AND LOCATIONS:
Overall Officials: AbdElKader A Hyder, MSc, Principal Investigator — Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Al-Azhar University; Wael A ElMohandes, PhD, Study Director — Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Al-Azhar University; Bahaa El-Din A Tawfik, PhD, Study Director — Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Al-Azhar University
Locations (1):
- Faculty of Dentistry, Al-Azhar University., Cairo, Egypt

REFERENCES:
- [Background] Krause M, Dorfler HM, Kruber D, Humpfner-Hierl H, Hierl T. Template-based temporomandibular joint puncturing and access in minimally invasive TMJ surgery (MITMJS) - a technical note and first clinical results. Head Face Med. 2019 Apr 2;15(1):10. doi: 10.1186/s13005-019-0194-8. PMID 30940211
- [Background] Steenks MH, Turp JC, de Wijer A. Reliability and Validity of the Diagnostic Criteria for Temporomandibular Disorders Axis I in Clinical and Research Settings: A Critical Appraisal. J Oral Facial Pain Headache. 2018 Winter;32(1):7-18. doi: 10.11607/ofph.1704. PMID 29370321
- [Background] Rani S, Pawah S, Gola S, Bakshi M. Analysis of Helkimo index for temporomandibular disorder diagnosis in the dental students of Faridabad city: A cross-sectional study. J Indian Prosthodont Soc. 2017 Jan-Mar;17(1):48-52. doi: 10.4103/0972-4052.194941. PMID 28216845